CLINICAL TRIAL: NCT05323526
Title: Validation of the Catquest-9SF Questionnaire in Greek Language
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES1/Th7/30-01-2020
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Cataract; Catquest-9SF
Keywords: cataract; catquest; validation; questionnaire; Rasch Analysis
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: 100 patients who will undergo cataract surgery
  Interventions: Diagnostic Test: Catquest-9SF questionnaire; Diagnostic Test: Demographics and clinical parameters

INTERVENTIONS:
Diagnostic Test: Catquest-9SF questionnaire — Patients complete the questionnaire preoperatively and postoperatively.
Diagnostic Test: Demographics and clinical parameters — The following clinical parameters are evaluated: age, gender, ocular and systemic comorbidities, educational level, preoperative and postoperative monocular distance uncorrected visual acuity (UVA), distance best spectacle-corrected visual acuity (BSCVA) of the eye for cataract surgery, binocular distance UVA and BSCVA, refraction, spherical equivalent (SE), and intraocular pressure.

SUMMARY:
Primary objective of this study is the validation of the Catquest-9SF questionnaire in the Greek population.

DETAILED DESCRIPTION:
The present study aims to validate the Catquest-9SF questionnaire in the Greek population. The Catquest-9SF is a questionnaire for assessing the quality of vision of patients with cataract. It consists of 9 questions, two of which concern the subjective assessment of the patient's vision and the other seven the patient's ability to perform various daily activities.

The Catquest-9SF questionnaire were translated into the Greek language by a translation team consisting of five members: one translation coordinator, two professional native English-speaking translators, one professional native Greek-speaking translator and one native Greek ophthalmologist fluent in English.

Patients participating in the study are asked to complete a questionnaire in Greek before and after cataract surgery. Upon completion of the data collection, data are processed and analyzed through Rasch analysis to determine whether the questionnaire can be used in clinical practice in this translated version.

The following clinical parameters are evaluated: age, gender, preoperative and postoperative monocular distance uncorrected visual acuity (UVA), distance best spectacle-corrected visual acuity (BSCVA) of the eye for cataract surgery, binocular distance UVA and BSCVA, refraction, spherical equivalent (SE), and intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral senile cataract with stage 2 nuclear opalescence according to the Lens Opacities Classification System III (LOCS-3) grading scale, and no severe cognitive impairment during their preoperative examination.

Exclusion Criteria:

* Patients with difficulty with the Greek language or dementia, Alzheimer's disease, severe stroke with mental disorder and conditions with the onset of mental retardation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cataract who will undergo cataract surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Rasch Analysis: Response category ordering | 3 months
  Response category ordering is evaluated graphically with category probability curves by observing whether the four response categories - omitting 'Cannot decide' as missing - (three category thresholds) are utilized in ascending order.
Rasch Analysis: Item fit statistics [infit and outfit mean square (MNSQ)] | 3 months
  Item fit statistics are used for the evaluation of the unidimensionality. When data fit well, the items should contribute to a single construct (visual disability) indicating the unidimensionality of the questionnaire (or the subscale). Both infit and outfit mean squares have an expected value of 1.0, with an ideal range of 0.7 to 1.3, and an acceptable range of 0.5 to 1.5) A value < 0.7 indicates too little variance and easily predicted questions, while > 1.3 indicates too much variance.
Rasch Analysis: Principal components analysis (PCA) | 3 months
  PCA is used for the evaluation of the unidimensionality. Two criteria are used; the PCA assessment is performed by comparing the amount of variance explained empirically and by the model, and the amount of variance explained by the first contrast (additional dimension). For unidimensionality, the unexplained variance in the first contrast of the residuals should be < 2.0 eigenvalue units, and ≥ 60% of variance should ideally be explained by the measure, while a percentage of ≥ 50% is acceptable.
Rasch Analysis: Person Separation Index (PSI) | 3 months
  PSI contributes to the assessment of the measurement precision of the Greek Catquest-9SF. PSI implies the questionnaire's ability to differentiate along its scale. The greater the value of person separation, the greater the questionnaire precision (acceptable person separation > 3.0).
Rasch Analysis: Person Reliability (PR) | 3 months
  PR contributes to the assessment of the measurement precision of the Greek Catquest-9SF. PR (ranging from 0 to 1) should be > 0.9 to be considered adequate, indicating a high ability to distinguish between the strata of person ability.
Rasch Analysis: Differential Item Functioning (DIF) | 3 months
  DIF indicates the differences between different subgroups of patients, since the questionnaire item calibration should be comparable across different patient groups. DIF occurs if patients from different subgroups with the same underlying true ability have an unequal probability of giving of a response to an item. DIF is assessed by evaluating age, gender, existence of ocular comorbidities, first vs second eye cataract surgery and binocular distance BSCVA. DIF of >1.0 logits is significant, DIF with values between 0.5 and 1.0 is minimal, and DIF <0.5 logits is considered absent.
Rasch Analysis: Τargeting | 3 months
  Τargeting of the questions to the patient sample, which indicates how well the items' difficulties match the person ability, is assessed to establish if the questions are appropriate for patients before and following cataract surgery. This can be assessed graphically by observing the spread along the person-item map and by the difference between the item and the person mean values. A well-targeted instrument requires the ability of the patients and the difficulty of the questions to be centered on the same mean (targeting of 0). In general, a mean difference in magnitude of ≥1 logit indicates significant mistargeting, while a difference of <1.0 logit indicates good targeting, with targeting of 0 being ideal. A positive value indicates that the items are too difficult relative to person's ability, while a negative value indicates that the items are too easy. A person-item map also visualizes the item hierarchy of difficulty, ranging from a minimum to maximum difficulty of performance.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (2):
- Greece (2):
  - Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros
  - General Hospital of Kalamata, Kalamata, Messinia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nanos P, Kouteliari V, Panagiotopoulou EK, Papadopoulos N, Ntonti P, Labiris G. Catquest-9SF questionnaire: Validation in a Greek-speaking population using Rasch analysis. PLoS One. 2022 Dec 7;17(12):e0278683. doi: 10.1371/journal.pone.0278683. eCollection 2022. PMID 36477289